CLINICAL TRIAL: NCT05484219
Title: Functional Navigation in Surgery of Cerebral Tumors and Vascular Malformations: a Prospective, Single Arm Clinical Trial
Brief Title: Functional Navigation in Surgery of Cerebral Tumors and Vascular Malformations
Acronym: FUN
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: technical issues
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Principal Investigator, Sklifosovsky Institute of Emergency Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9f
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tumor, Brain; Arteriovenous Malformations; Cavernoma
Keywords: brain tumor; arteriovenous malformation; cavernoma; cavernous malformation; functional navigation
MeSH Terms: conditions — Brain Neoplasms; Arteriovenous Malformations; Hemangioma, Capillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery (Experimental): Image-guided resection of brain tumors and vascular malformations
  Interventions: Device: Functional navigation

INTERVENTIONS:
Device: Functional navigation — Surgeon removes brain tumor or vascular malformation and assesses location of motor areas with functional navigation and intraoperative neuromonitoring

SUMMARY:
The purpose of the study is to assess accuracy, advantages of functional neuronavigation and calculate safe distance from motor areas to brain tumors and vascular malformations in image-guided surgery.

DETAILED DESCRIPTION:
Functional images (functional magnetic resonance imaging (fMRI), transcranial magnetic stimulation (TMS), tractography) loaded in neuronavigation are called functional navigation. It is usually combined with anatomical data and allows to display eloquent brain areas. Currently there are plenty of studies concerning possibilities of it's use. In our research we plan to confirm this data and to supplement them with calculating a safe distance from motor areas to various mass lesions in preoperative scans where neurological deficits is not likely to appear after surgery. In case of success this data can be a foundation for further researches specifying indications for use of intraoperative neuromonitoring and possibility of it's replacement with functional navigation in some cases.

The purpose of the study is to assess accuracy, advantages of functional neuronavigation and calculate safe distance from motor areas to brain tumors and vascular malformations in image-guided surgery. For each patient a surgeon intraoperatively will assess locations of motor cortex and corticospinal tract found with direct cortical and subcortical stimulation and capture them. After surgery he will compare this data with functional preoperative scans and virtual motor centers constructed based on tractography. Influence of various factors on precision of functional navigation will be studied and safe distance between motor brain areas and mass lesion borders will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* all intracranial tumors
* arteriovenous malformations
* cavernous malformations
* supratentorial localization
* newly diagnosed
* age 18-79 years
* unaltered consciousness
* error of patient registration in neuronavigation no more than 2 mm
* possibility to perform "positive mapping" strategy

Exclusion Criteria:

* contraindications to magnetic resonance imaging or transcranial magnetic stimulation
* inability to build tractography in neuronavigation
* predicting of intraoperative brain shift 6 mm and more without possibility to correct it
* real intraoperative brain shift 6 mm and more without possibility to correct it
* previously performed brain radiotherapy
* pregnancy
* breast feeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of functional navigation (in millimeters) | Intraoperatively
  Maximal distance from the most remote margin of cortical hand/leg motor area or corticospinal tract in the area of corona radiata in functional navigation to the nearest margin of this area/tract in direct cortical/subcortical stimulation
Accuracy of location of cortical hand/leg motor area, built according to tractography (in millimeters) | Intraoperatively
  Maximal distance from the most remote margin of cortical hand/leg motor area, built according to tractography and loaded into navigation, to the nearest margin of this area in direct cortical stimulation

SECONDARY OUTCOMES:
Constancy of location of cortical hand/leg motor area in fMRI/TMS in relation to precentral gyrus (in millimeters) | Within 2 days before surgery
  Maximal distance from the most remote margin of cortical hand/leg motor area in fMRI/TMS to the nearest margin of precentral gyrus
Factors, violating precision of fMRI/TMS/tractography | Within 2 days before surgery
  Which factors lead to disappearing, thinning and dislocation of cortical hand/leg motor areas and corticospinal tract in fMRI/TMS/tractography
Motor function (in grades) | Within 10 days after surgery
  Motor function is assessed in Medical Research Council scale
Distance to stop resection border (in millimeters) | Intraoperatively
  Minimal distance from the nearest margin of cortical hand/leg motor area or corticospinal tract to the nearest border of resection of tumor/vascular malformation
Safe resection distance in functional navigation (in millimeters) | Within 10 days after surgery
  This outcome is only measured in patients with no deterioration of motor function after surgery. Safe resection distance = accuracy of functional navigation + distance to stop resection border
Duration of direct cortical and subcortical mapping (in minutes) | Intraoperatively
  How long did it take to perform direct cortical and subcortical mapping
Extent of resection (in percents) | Within 48 hours after surgery
  Extent of resection = (preoperative tumor volume - postoperative tumor volume) / preoperative tumor volume x 100
Karnofsky performance status (in percents) | Within 10 days after surgery
  Assessment of patients' possibilities to self-service in Karnofsky Performance Status scale
Cerebral complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which cerebral complications arose after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No